CLINICAL TRIAL: NCT06346912
Title: A Study of CD19-BAFF CAR-T Cells Therapy for Patients With Relapsed and/or Refractory B-cell ALL and B-cell NHL
Brief Title: CD19-BAFF CAR-T Cells Therapy for Patients With Relapsed / Refractory B-cell ALL and B-cell NHL
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2023022
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-12

CONDITIONS: Acute Lymphoblastic Leukemia,B-Cell; Non-hodgkin Lymphoma,B Cell
Keywords: CD19-BAFF CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CD19-BAFF Targeted CAR T-cells (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CD19-BAFF Targeted CAR T-cells

INTERVENTIONS:
Biological: CD19-BAFF Targeted CAR T-cells — Each subject receive CD19-BAFF Targeted CAR T-cells by intravenous infusion
  Other Names: CD19-BAFF Targeted CAR T-cells injection

SUMMARY:
Clinical Trial for the safety and efficacy of CD19-BAFF CAR-T cells therapy for refractory/relapsed B-cell acute lymphoblastic leukemia and B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
In this study, 20 patients with relapsed refractory B-cell ALL and B-cell NHL were proposed to undergo CD19-BAFF CAR-T cell therapy. Under the premise that its safety has been clarified in previous studies, further observation and evaluation of the effectiveness of CD19-BAFF CAR-T cell therapy for relapsed refractory B-cell ALL and B-cell NHL; At the same time, on the basis of expanding the sample size, more safety data on CD19-BAFF CAR-T cell treatment for relapsed refractory B-cell ALL and B-cell NHL were accumulated, including rare and delayed complications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Gender unlimited，18< Age;
* 2. Patients diagnosed with B-cell acute lymphoblastic leukemia through histological or immunophenotyping tests; The clear diagnosis of B-cell non Hodgkin's lymphoma by cellular or histopathological examination mainly includes diffuse large B-cell lymphoma, follicular lymphoma, and mantle cell lymphoma
* 3. Relapsed or refractory CD19+ B-ALL (meeting one of the following conditions):

  1. CR not achieved after standardized chemotherapy;
  2. CR achieved following the first induction, but CR duration is less than 12 months;
  3. Ineffectively after first or multiple remedial treatments;
  4. 2 or more relapses;
* 4. The number of primordial cells (lymphoblast and prolymphocyte) in bone marrow is >5% (by morphology), and/or >1% (by flow cytometry);
* 5. Philadelphia-chromosome-negative (Ph-) patients; or Philadelphia-chromosome-positive (Ph+) patients who cannot tolerate TKI treatments or do not respond to 2 TKI treatments;
* 6. Relapsed or refractory B-NHL (meeting one of the following conditions):

  1. No response or relapse after second-line or above chemotherapy regimens;
  2. Primary drug resistance;
  3. Relapse after auto-HSCT;
* 7. At least one assessable tumor lesion per Lugano 2014 criteria;
* 8. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
* 9. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
* 10. No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
* 11. Estimated survival time ≥ 3 months;
* 12. ECOG performance status 0 to 2;
* 13. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

* 1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
* 2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
* 3. Pregnant/lactating women, or male or female patients with fertility who are unwilling to take effective contraceptive measures during the study period or at least 6 months after the last cell infusion
* 4. Patients with HIV infection;
* 5. Active infection of hepatitis B virus or hepatitis C virus;
* 6. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 7. Other uncontrolled diseases that were not suitable for this trial;
* 8. Individuals who have received CAR-T therapy, CAR-NK therapy, or any other gene modified cell therapy product within 6 months;
* 9. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 years after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Overall response rate ,ORR | Up to 12 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Duration of remission ,DOR | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Event-free survival, EFS | Up to 1 years after CAR-T infusion
  The time from first achieving CR/CRi to relapse or death
Overall survival, OS | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China